CLINICAL TRIAL: NCT05511883
Title: Periosteal Chondrosarcoma: a Single Institution Experience
Acronym: PC
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Alberto Righi, MD, PhD, Istituto Ortopedico Rizzoli
Other Study IDs: 136/2020
Record Dates: First submitted 2021-09-21; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-09

CONDITIONS: Periosteal Chondrosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periosteal chondrosarcoma is a low-grade, malignant cartilaginous bone neoplasm that arises on the surface of bone, predominantly in the metaphysis of long bones.

Periosteal chondrosarcoma is an infrequent chondrosarcoma subtype which accounts for less than 1% of all chondrosarcomas (1) and has a peak incidence in the fourth decade (2).

It has a reported incidence of local recurrences of 13-28% and a low metastatic potential, with distant recurrences occurring mostly in lungs (3).

Contrary to conventional chondrosarcomas, grading of periosteal chondrosarcomas seems not to predict prognosis. IDH1 and IDH2 mutations, characteristics of central chondromas/chondrosarcomas, have been also found in a subset of periosteal chondrosarcomas (1, 4).

These observations are based on the results from smaller series of cases (1, 5, 6), although the impact of histopathological characteristics on survival, local recurrence and metastases should be assessed in larger series of cases.

The aim of the present study is to review all the cases with a diagnosis of primary periosteal chondrosarcoma treated at the Rizzoli Institute from 1900 up to 31 December 2019, retrospectively.

The study will exam all the clinical, radiological, and histological features of this tumor with regard importance of medullary involvement, the IDH1/2 gene status, the types of treatment, the status of surgical margins, the presence of progression (dedifferentiation) areas and the relationship of these factors to individual outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Institute from 01 Jan 1900 to 31 Dec 2019
* Diagnosis of peristeal chondrosarcoma
* Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

* Patients with histological diagnosis different from periosteal chondrosarcoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients considered eligible will be included in the study, after providing a written informed consent.
  Since we will include cases of several decades ago, and due to the high incidence of mortality of the disease under investigation, it would be possible that some eligible subjects will be deceased.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Periosteal Chondrosarcoma: a single institution experience | act baseline
  the IDH1/2 gene status.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided